CLINICAL TRIAL: NCT00463476
Title: Assessment of the Immunogenicity and Safety of Japanese Encephalitis Live Attenuated SA 14-14-2 Vaccine in Children in Sri Lanka
Brief Title: Boosterability of Live Attenuated Japanese Encephalitis (JE) Vaccine in Children Who Have Previously Received Inactivated JE Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PATH (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: JEV04
Record Dates: First submitted 2007-04-18; First posted 2007-04-20 (Estimated); Results first posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2018-09

CONDITIONS: Japanese Encephalitis
MeSH Terms: conditions — Encephalitis, Japanese

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2-year olds (Experimental): Healthy children 2 years of age (±3 months) who had previously received all vaccinations recommended under the Sri Lankan childhood immunization schedule according to their age. Subjects must have previously received inactivated mouse brain-derived Japanese Encephalitis vaccine (IMBV) at the recommended 12 and 13 months of age. Subjects received one dose of Live, Attenuated Japanese Encephalitis SA 14-14-2 Vaccine (LJEV).
  Interventions: Biological: Live, Attenuated Japanese Encephalitis SA 14-14-2 Vaccine (LJEV)
- 5-year olds (Experimental): Healthy children 5 years of age (±3 months) that met all other eligibility criteria. Subjects must have previously received inactivated mouse brain-derived Japanese Encephalitis vaccine (IMBV) at the recommended 12, 13, and 24 months of age. Subjects received one dose of Live, Attenuated Japanese Encephalitis SA 14-14-2 Vaccine (LJEV).
  Interventions: Biological: Live, Attenuated Japanese Encephalitis SA 14-14-2 Vaccine (LJEV)

INTERVENTIONS:
Biological: Live, Attenuated Japanese Encephalitis SA 14-14-2 Vaccine (LJEV) — Manufactured by Chengdu Institute of Biological Products (CDIBP), Chengdu, China; batch 200611A078-1. Administered subcutaneously in the right upper arm using 23 gauge needles.

SUMMARY:
To facilitate introduction of live attenuated SA 14-14-2 Japanese encephalitis vaccine (LJEV) into the National Immunization Programme of Sri Lanka, we evaluated the safety and immunogenicity of co-administration of LJEV and measles vaccine in children at 2 and 5 years of age. The primary hypothesis was that the seropositivity rate at 28 days post vaccination of SA 14-14-2 in subjects 2 and 5 years of age who have already received at least two doses of mouse brain-derived inactivated JE vaccine is greater than 80%.

Japanese encephalitis virus is the leading cause of viral neurological disease and disability in Asia. The severity of sequelae, together with the volume of cases, make JE the most important cause of viral encephalitis in the world. Approximately 3 billion people-including 700 million children-live in areas at risk in Asia for JE. JE most commonly infects children between the ages of 1 and 15 years, and can also infect adults in areas where the virus is newly introduced. More than 50,000 cases are reported annually and cause an estimated 10,000 to 15,000 deaths. This figure is believed to represent only a small proportion of the disease burden that actually exists.

DETAILED DESCRIPTION:
JE virus is an arbovirus that causes a devastating neurological disease resulting in high rates of mortality or neurologic sequelae. The severity of sequelae, together with the volume of cases, makes JE an important cause of encephalitis. The disease is endemic across temperate and tropical zones of Asia,and because of its zoonotic cycle, eradicating JE from the environment is unrealistic. Universal childhood vaccination is essential for disease control.

Concern in Japan over a rare but potentially dangerous adverse event associated with a mouse brain-derived vaccine led the manufacturer in Japan to discontinue production in 2005, thus limiting global supply of inactivated JE vaccines and raising costs for remaining inactivated vaccines. In August of 2006, the World Health Organization stated in its position paper on Japanese encephalitis vaccines that the mouse brain-derived vaccine should be replaced by a new generation of JE vaccines.

In Sri Lanka, immunization against JE began in 1988. By 2006, two types of JE vaccines were available for use in Sri Lanka-inactivated mouse brain-derived vaccine and live attenuated SA-14-14-2 JE vaccine (LJEV). Only the inactivated vaccine was being used in the country's public-sector immunization program. It is given to children in 3 doses, at 12 months of age, 13 months of age, and 2 years of age. A booster dose must also be given to children at 5 years of age. If Sri Lanka decides to replace the inactivated JE vaccine with the live attenuated JE vaccine, there will be many children who still need a 3rd or booster dose of the inactivated JE vaccine. This research study was done to see if the live attenuated vaccine would work well to replace the inactivated JE vaccine and if it is safe in Sri Lankan children. The study was conducted in three peri-urban health divisions of low JE endemicity in the District of Colombo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy child 2 years (±3 months) or 5 years (±3 months) of age at the enrollment visit.
* Subject was a full-term infant.
* Subject's parent or legal guardian is literate and willing to provide written informed consent.
* Subject is up-to-date for all vaccinations recommended in the Sri Lankan childhood immunization schedule.

Exclusion Criteria:

* Enrolled in another clinical trial involving any therapy.
* Subject and/or parent(s) or guardian(s) are unable to attend the scheduled visits or comply with the study procedures.
* Received any non-study vaccine within 2 weeks prior to enrolment or refusal to postpone receipt of such vaccines until 28 days after study entry.
* Prior or anticipated receipt of immune globulin or other blood products, or injected or oral corticosteroids or other immune modulator therapy except routine vaccines within 6 weeks of administration of study vaccine. Individuals on a tapering dose schedule of oral steroids lasting <7 days may be included in the trial as long as they have not received more than one course within the last 2 weeks prior to enrolment.
* History of documented or suspected encephalitis, encephalopathy, or meningitis.
* History of measles.
* History of Japanese encephalitis.
* Serious adverse event related (i.e., possible, probably, definite) to previous receipt of any JE vaccine, if applicable.
* Persistent inconsolable crying (>3 hours) observed after previous receipt of any JE vaccine, if applicable.
* Hypotonic - hyporesponsiveness after past receipt of any JE vaccine, if applicable.
* Suspected or known hypersensitivity to any of the investigational or marketed vaccine components.
* History of serious chronic disease (cardiac, renal, neurologic, metabolic, or rheumatologic).
* Underlying medical condition such as inborn errors of metabolism, failure to thrive, bronchopulmonary dysplasia, or any major congenital abnormalities requiring surgery or chronic treatment.
* History of thrombocytopenic purpura.
* History of seizures, including history of febrile seizures, or any other neurologic disorder.
* Known or suspected immunologic function impairment of any kind and/or known HIV infection.
* Parent with known or suspected immunologic function impairment of any kind and/or known HIV infection.
* Any condition that, in the opinion of the investigator, would pose a health risk to the participant or interfere with the evaluation of the study objectives.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 305 (Actual)
Dates: Start 2007-07-09 (Actual); Primary Completion 2007-11-01 (Actual); Study Completion 2008-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nihal Abeysinghe, MD, MSc, Principal Investigator — Epidemiological Unit, Sri Lanka Ministry of Healthcare and Nutrition
Locations (3):
- Sri Lanka (3):
  - Homagama MOH Division Medical Office, Homagama, District of Colombo
  - Kolonnawa MOH Division Medical Office, Kolonnawa, District of Colombo
  - Moratuwa MOH Division Medical Office, Moratuwa, District of Colombo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy children 2 and 5 years of age who had previously received two and three doses of inactivated mouse brain-derived vaccine (IMBV), respectively, were enrolled in the Colombo District of Sri Lanka between July and October 2007.
Groups:
- 2-year Olds: Healthy children 2 years of age who had previously received IMBV at the recommended 12 and 13 months of age received one dose of live, attenuated Japanese encephalitis SA 14-14-2 vaccine (LJEV) administered subcutaneously in the right upper arm on Study Day 0.
- 5-year Olds: Healthy children 5 years of age who had received IMBV at the recommended 12, 13, and 24 months of age received one dose of live, attenuated Japanese encephalitis SA 14-14-2 vaccine (LJEV) administered subcutaneously in the right upper arm on Study Day 0.
Period: Overall Study
Arm/Group | 2-year Olds | 5-year Olds
Started | 151 | 154
Completed | 149 | 151
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2-year Olds | 5-year Olds | Total
Number analyzed (Participants) | 151 | 154 | 305
Age, Continuous [Mean (Standard Deviation); unit: months] | 24.5 (1.4) | 60.4 (1.6) | 42.6 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 78 | 150
  Male | 79 | 76 | 155
Region of Enrollment [Number; unit: participants]
  Sri Lanka | 151 | 154 | 305

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Demonstrated Seropositivity for Japanese Encephalitis (JE) Neutralizing Antibodies
Description: Blood serum was collected immediately before administration (Day 0), Day 28, and 1 year later. Serum neutralizing antibodies to the Beijing-1 JE strain were measured by plaque reduction neutralization test (PRNT) where the neutralizing titer was measured as the inverse dilution at which plaque counts were reduced by 50%. Seropositivity was defined as a titer of ≥ 1:10.
Time Frame: Day 0 (pre-vaccination) and 28 days and 1 year post-vaccination
Population: The per-protocol analysis set included all participants of the appropriate age at study entry (2 years of age ±3 months and 5 years of age ±3 months for each group respectively) who received LJEV at Day 0 and with valid serology laboratory results 28 days post-vaccination. Five participants did not complete the 1-year post-vaccination visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2-year Olds | 5-year Olds
Number analyzed (Participants) | 147 | 147
percentage of participants
  Day 0 | 98.0 [94.2 to 99.6] | 99.3 [96.3 to 100.0]
  Day 28 | 100.0 [97.5 to 100.0] | 100.0 [97.5 to 100.0]
  One year: number analyzed (Participants) | 145 | 144
  One year | 100.0 [97.5 to 100.0] | 99.3 [96.2 to 100.00]

2. Secondary Outcome: Geometric Mean Titer (GMT) of Japanese Encephalitis (JE) Neutralizing Antibodies
Description: Blood serum was collected immediately before administration (Day 0), Day 28, and 1 year later. Serum neutralizing antibodies to the Beijing-1 JE strain were measured by plaque reduction neutralization test (PRNT) where the neutralizing titer was measured as the inverse dilution at which plaque counts were reduced by 50%.
Time Frame: Day 0 and 28 days and 1 year post-vaccination
Population: Per-protocol analysis set; 5 participants did not complete the 1-year post-vaccination visit.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 2-year Olds | 5-year Olds
Number analyzed (Participants) | 147 | 147
titer
  Day 0 | 697 [551 to 883] | 926 [733 to 1170]
  Day 28 | 3175 [2744 to 3672] | 2776 [2400 to 3210]
  1 year: number analyzed (Participants) | 145 | 144
  1 year | 3170 [2674 to 3758] | 2585 [2131 to 3136]

3. Secondary Outcome: Number of Participants With Immediate Reactions, Local and Systemic Reactions, and Unsolicited Adverse Events (AE)
Description: Participants were monitored for immediate AEs and local reactions for 30 minutes after each injection by a study physician. Thereafter, parents recorded axillary temperature, local reactions (redness, swelling, pain, and other local reactions), and systemic symptoms (high-grade fever, anorexia, crying, diarrhea, drowsiness, insomnia, irritability, vomiting, and other systemic symptoms) in a study diary for 7 days afterwards. Study staff called the participants' parents 2 days after vaccination and monthly through 1 year to inquire about the child's well being and review the diary card. The participant was visited at home on Day 7 to review and collect the reactogenicity diary card. The participant returned to the vaccination clinic on Day 28, 6 months, and 1 year to be examined, have a blood draw, and review any AEs or serious adverse events (SAE) with parents.
Time Frame: Day 0 and 28 days and 1 year post-vaccination
Population: All enrolled participants who received at least one dose of the live JE vaccine. Not all participants were followed for a full 30 minutes after injection.
Measure: Count of Participants; unit: Participants
Arm/Group | 2-year Olds | 5-year Olds
Number analyzed (Participants) | 151 | 154
Participants
  Immediate reactions within 30 minutes: number analyzed (Participants) | 148 | 144
  Immediate reactions within 30 minutes | 0 | 1
  Solicited local reactions Days 0-3 | 31 | 46
  Solicited local reactions Days 4-7 | 1 | 6
  Solicited systemic reactions Days 0-7 | 44 | 38
  Solicited systemic reactions > 7 days | 12 | 5
  Unsolicited systemic reactions Days 0-7 | 15 | 15
  Unsolicited systemic reactions > 7 days | 11 | 12
  Any non-serious adverse events Days 8-28 | 54 | 54
  Related adverse events at any time | 0 | 1
  Serious adverse events, Days 8-365 | 22 | 8

4. Secondary Outcome: Number of Participants Experiencing Solicited Local Reactions Up to 3 Days Post-vaccination
Description: Parents recorded local reactions (redness, swelling, pain, and other local reactions) in a study diary.
  Events were assessed by the clinician to quantify intensity using the following guidelines:
  * Mild: Events required minimal or no treatment and do not interfere with the child's functioning.
  * Moderate: Events resulted in a low level of concern with therapeutic measures. Moderate events may cause some interference with functioning.
  * Severe: Events interrupted the child's functioning and may have required systemic drug therapy or other treatment. Severe events are usually incapacitating.
Time Frame: 3 days post-vaccination
Population: All enrolled participants who received at least one dose of the live JE vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | 2-year Olds | 5-year Olds
Number analyzed (Participants) | 151 | 154
Participants
  Any local reactions | 31 | 46
  Mild local reactions | 27 | 41
  Moderate local reactions | 4 | 5
  Severe local reactions | 0 | 0
  Redness (Erythema) | 7 | 7
  Pain | 28 | 44
  Swelling | 8 | 9

5. Secondary Outcome: Number of Participants Experiencing Solicited Systemic Reactions up to 7 Days Post-vaccination
Description: Parents recorded axillary temperature and systemic symptoms (high-grade fever, anorexia, crying, diarrhea, drowsiness, insomnia, irritability, vomiting, and other systemic symptoms) in a study diary for 7 days after vaccination. The participant was visited at home on Day 7 to review and collect the reactogenicity diary card.
  Events were assessed by the clinician to quantify intensity using the following guidelines:
  * Mild: Events required minimal or no treatment and do not interfere with the child's functioning.
  * Moderate: Events resulted in a low level of concern with therapeutic measures. Moderate events may cause some interference with functioning.
  * Severe: Events interrupted the child's functioning and may have required systemic drug therapy or other treatment. Severe events are usually incapacitating.
Time Frame: 7 days post-vaccination
Population: All enrolled participants who received at least one dose of the live JE vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | 2-year Olds | 5-year Olds
Number analyzed (Participants) | 151 | 154
Participants
  Any systemic reaction | 44 | 38
  Severe systemic reaction | 1 | 1
  Fever: Any severity | 12 | 16
  Fever: Severe | 0 | 0
  Anorexia: Any severity | 28 | 16
  Anorexia: Severe | 0 | 1
  Crying: Any severity | 15 | 8
  Crying: Severe | 0 | 0
  Diarrhea: any severity | 0 | 1
  Diarrhea: Severe | 0 | 1
  Tiredness: Any | 9 | 5
  Tiredness: Severe | 0 | 0
  Insomnia: Any severity | 13 | 5
  Insomnia: Severe | 0 | 0
  Irritability: Any severity | 6 | 5
  Irritability: Severe | 1 | 0
  Vomiting: Any severity | 6 | 6
  Vomiting: Severe | 0 | 0

6. Post Hoc Outcome: Number of Participants With Baseline Japanese Encephalitis (JE) Neutralizing Antibodies ≥ 10 Experiencing Fold-level Increases in JE Neutralizing Antibodies From Pre-vaccination to 28 Days Post-vaccination
Description: Compares geometric mean titers (GMT) for baseline and 28 days post-vaccination among participants seropositive for neutralizing antibodies against JE virus (titer of ≥1:10) at Baseline. Serum neutralizing antibodies to the Beijing-1 JE strain were measured by plaque reduction neutralization test (PRNT) where the neutralizing titer was measured as the inverse dilution at which plaque counts were reduced by 50%.
Time Frame: Baseline (Day 0) and 28 days post-vaccination
Population: Per-protocol analysis set with baseline Japanese encephalitis (JE) neutralizing antibodies ≥ 10.
Measure: Count of Participants; unit: Participants
Arm/Group | 2-year Olds | 5-year Olds
Number analyzed (Participants) | 144 | 146
Participants
  < 2.00-fold increase | 42 | 63
  2.00-2.99-fold increase | 12 | 15
  3.00-3.99-fold increase | 14 | 9
  ≥ 4.00-fold increase | 76 | 59

ADVERSE EVENTS:
Time Frame: 1 year for serious adverse events, 28 days for non-serious adverse events.
Arm/Group | 2-year Olds | 5-year Olds
All-Cause Mortality (participants affected / at risk) | 0/151 | 0/154
Serious Adverse Events (participants affected / at risk) | 22/151 | 8/154
Other Adverse Events (participants affected / at risk) | 54/151 | 54/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2-year Olds (N=151) | 5-year Olds (N=154)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Enterobiasis (Infections and infestations) | 0 (0) | 1 (1)
Gastritis viral (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 5 (8) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Viral infection (Infections and infestations) | 7 (7) | 1 (1)
Accidental exposure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tongue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Febrile convulsion (Nervous system disorders) | 2 (3) | 0 (0)
Penile swelling (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2-year Olds (N=151) | 5-year Olds (N=154)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 16 (16) | 17 (17)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Enterobiasis (Infections and infestations) | 0 (0) | 1 (1)
Gastritis viral (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 5 (6) | 3 (3)
Nasopharyngitis (Infections and infestations) | 17 (17) | 11 (11)
Rash pustular (Infections and infestations) | 0 (0) | 4 (4)
Respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 7 (7) | 1 (1)
Accidental exposure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cephalhaematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tongue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Febrile convulsion (Nervous system disorders) | 2 (2) | 0 (0)
Penile swelling (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (20) | 20 (20)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No